CLINICAL TRIAL: NCT07142005
Title: Cultural Adaptation of an Educational Tool in Medullary Thyroid Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0198; NCI-2025-04498 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-06-20; First posted 2025-08-26 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-06

CONDITIONS: Medullary Thyroid Cancer (MTC); Cultural Adaptation
MeSH Terms: conditions — Carcinoma, Medullary | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interviews — * Questionnaires/Survey Measures
  * Qualitative Instruments

SUMMARY:
To find good information about medullary thyroid cancer that is easy to understand and reliable, so researchers aim to design some new educational materials to help.

DETAILED DESCRIPTION:
Primary Objectives

1. To co-develop a culturally-adapted educational tool for the Latino/Latina MTC population using the previously developed MTCEducate.org as a framework. (Phase 1)
2. To test, refine, and produce a culturally adapted educational prototype and is intended to assess participants' understanding after reviewing the decision aid as part of the iterative testing and refinement process (Phase 2)

Secondary Objectives

1. To assess the tool's acceptability post-production among a broader population of Latino(a) MTC participants and caregivers using the Ottawa Acceptability Scale (Phase 3)
2. To disseminate the educational tool to a broader population of Latino(a)s
3. To summarize the clinico-demographics of educational tool users

ELIGIBILITY:
Inclusion criteria:

* Provision of signed and dated informed consent form
* Males and females; Age: ≥18 years old
* Identified ethnicity as "Hispanic" or "Latino/Latina"
* Ability to read, write, and speak Spanish
* Those who are pregnant are eligible to participate
* Have or will face this decision, including: a. Participant/survivor - who has medullary thyroid carcinoma, as determined by a clinician or documented in Multi-Institutional Medullary Thyroid Cancer Collaborative Registry; b. Caregiver/family member - of Participant/survivor who has medullary thyroid carcinoma, as nominated by the Participant/survivor

Exclusion Criteria:

* Those < age 18
* Ethnic identity as non-Hispanic or non-Latino/a individual
* Individuals with cognitive or psychological impairment (e.g., depression, anxiety, severe mental illness as documented in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaires/Survey Measures | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Grubbs, MD, Principal Investigator — eggrubbs@mdanderson.org
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org